CLINICAL TRIAL: NCT06371950
Title: Gut Microbiome in Orthopaedics: Effect of Probiotics on Initial Implant Migration and Joint Inflammation After Total Knee Replacement
Brief Title: Gut Microbiome in Orthopaedics
Acronym: GUMBO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to secure regulatory documentation for probiotic
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Brent Lanting, Orthopaedic surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 123608
Record Dates: First submitted 2024-02-27; First posted 2024-04-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Total Knee Arthroplasty; Inflammation; Gastrointestinal Health
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic DE111® (Experimental): 1 capsule of probiotic DE111® containing 5 billion CFU Bacillus subtilis, to be taken once daily starting 3 weeks prior to surgery until 6 weeks after surgery.
  Interventions: Dietary Supplement: Probiotic Formula Bacillus subtilis
- Placebo (Placebo Comparator): 1 capsule of placebo, to be taken once daily starting 3 weeks prior to surgery until 6 weeks after surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Formula Bacillus subtilis — 5 billion colony forming units (CFU) per day for 9 weeks (3 weeks before surgery to six weeks after surgery)
  Other Names: DE111®
  Arms: Probiotic DE111®
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Patients having knee replacement surgery regularly experience joint pain and compromised bone quality leading to implant loosening and periprosthetic fractures. The role of the gut microbiome, which is the collection of bacteria and other microbes within the human gastrointestinal tract, is just beginning to be recognized, including its potential effects on pain, infection, and loosening after total joint replacement. Antibiotics are regularly used in orthopaedic surgery to reduce the risk of infection, but they also harm gut microbiota and reduce their potentially beneficial effects. Probiotics may have a role to play in enhancing bone quality and decreasing synovial inflammation after joint replacement surgery, and this study will explore the potential relationship of probiotic use with implant migration, bone density, and patient outcomes.

This study is a randomized, controlled, double-blinded trial comparing probiotic use with placebo in post-menopausal women undergoing primary total knee replacement. The main questions it aims to answer are:

* to compare implant migration between groups from baseline to six weeks post-surgery
* to compare bone density and joint inflammation between groups from baseline to six weeks post-surgery
* to compare gut microbiome composition and patient-reported outcome measures between groups from baseline to six weeks post-surgery

DETAILED DESCRIPTION:
Participants will take a daily probiotic (DE111®) or placebo once daily starting 3 weeks prior to surgery until six weeks after surgery. The following will be completed at baseline and 6 weeks:

* Bloodwork
* Fecal sample collection
* MRSA swab
* Patient-reported outcome measures
* CT imaging scan

In addition, the following will be done:

* Intraoperative fluid and tissue collection
* Positron Emission Tomography-Magnetic Resonance Imaging (PET-MRI) scan at 6 weeks post-surgery

Researchers will compare the probiotic and placebo groups for any significant differences in implant stability, bone quality, inflammation, gut microbiome composition, and pain.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to any study-related activities
* Postmenopausal female patients of London Health Sciences Centre (LHSC) aged 55-75 years
* Scheduled to undergo primary total knee replacement for osteoarthritis

Exclusion Criteria:

* Unable to understand and respond to the provided questionnaires
* Male sex
* Inflammatory arthritis
* Periprosthetic infection
* Prior surgery with hardware insertion in the target knee
* Metabolic syndrome
* Inflammatory bowel disease
* Body mass index <18.5 kg/m2
* Immune-compromised condition (e.g. AIDS, lymphoma, patients undergoing long-term corticosteroid treatment)
* Any contraindications for PET-MRI
* Allergy to cephalosporin antibiotics

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Implant Migration | baseline, 6 weeks
  Tibial component migration over time calculated by measuring the position of the component compared to the bone using CT imaging.

SECONDARY OUTCOMES:
Bone Density | baseline, 6 weeks
  Volumetric bone mineral density over time measured in the anteromedial, anterolateral, posteromedial, and posterolateral regions surrounding the tibial component using CT imaging.
Magnitude of 18-F-Fluoroethyl(2-(2-fluoroethoxy)phenyl)-proprionate ([¹⁸F]FEPPA) Tracer Uptake | 6 weeks
  Magnitude of standardized uptake values (SUV) of the [¹⁸F]FEPPA tracer uptake in the synovium as measured by PET-MRI. SUV will be calculated using the mean signal intensity, body weight, and decay-corrected injected dose.

OTHER OUTCOMES:
Veterans Rand 12-Item Health Survey (VR-12) | pre-operative, 6 weeks
  Patient-reported outcome measure observing physical and mental health status of patient. Contains 12 questions about 8 health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. For each domain, the scores range from 0 to 100, with higher scores indicating better health-related quality of life. The minimum score is 0, indicating the lowest level of health or well-being, and the maximum score is 100, indicating the highest level of health or well-being.
EuroQol-5D (EQ-5D) | pre-operative, 6 weeks
  Patient-reported outcome measure to assess quality of life on a scale of 0 (worst) to 100 (best). Higher scores indicate better quality of life.
Western Ontario McMaster Osteoarthritis Index (WOMAC) | pre-operative, 6 weeks
  Patient-reported outcome measure to assess function, pain and stiffness on a scale of 0 (better function/pain/stiffness) to 100 (worse function/pain/stiffness). Higher scores indicate worse pain, stiffness, and functional limitations.
Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP) | pre-operative, 6 weeks
  Patient-reported questionnaire to assess experience with constant and intermittent pain on a scale of 0 (no pain) to 4 (extreme pain). A higher score indicates worse pain.
Patient Global Assessment (PGA) | pre-operative, 6 weeks
  Patient-reported scale question to measure global disease activity on a range of 0 (doing very well) to 10 (doing very poorly). A higher score indicates worse condition.
University of California, Los Angeles (UCLA) Activity Score | pre-operative, 6 weeks
  Patient-reported outcome measure assessing activity level of patient. Contains a 10-level scale with 1 representing a patient who is inactive and dependent on others, to 10 representing a patient who regularly participates in impact sports. A higher score indicates a greater activity level.
Oxford Knee Score - English for Canada | pre-operative, 6 weeks
  Patient-reported outcome measure to assess level of function, activities of daily living, and effects of pain over preceding four weeks, measured with 12 questions each on a scale from 0 (worst outcome) to 4 (best outcome). A higher score represents a better outcome, with total score range from 0-48
Knee Society Score (KSS) | pre-operative, 6 weeks
  Functional outcome measure. Contains 5 sections measuring patient symptoms (none to severe), satisfaction (very satisfied to very dissatisfied), expectation (too high to too low), functional activities, and discretionary knee activities. Functional activities are split into walking and standing (with or without aids and the duration), standard activities (no bother to cannot do), and advanced activities (no bother to cannot do). Discretionary knee activities measure difficulty with the three most important activities for the patient (no bother to cannot do). Higher scores indicate greater patient outcomes.
Presence of MRSA | pre-operative, 6 weeks
  Participants will provide a Methicillin-Resistant Staphylococcus Aureus (MRSA) swab sample. Presence of MRSA will be compared over time and between groups.
Microbial Diversity - Taxonomic Differences | pre-operative, 6 weeks
  Participants will provide a fecal sample. Microbial DNA will be extracted from the samples for 16S ribosomal ribonucleic acid (rRNA) sequencing so taxonomy can be assigned. The Shannon index for microbial diversity will be calculated and used to determine taxonomic differences in composition and diversity within and between samples.
Microbial Diversity - Taxonomic Correlation | pre-operative, 6 weeks
  Participants will provide a fecal sample. Microbial DNA will be extracted from the samples for 16S ribosomal ribonucleic acid (rRNA) sequencing so taxonomy can be assigned. Taxonomic correlations to other clinical and metadata in the study will be determined.
Diet and Supplement Questionnaire | pre-operative
  Patient-reported questionnaire collecting probiotic and supplement consumption habits and gastrointestinal symptoms. Consumption of fermented foods or drinks containing live bacteria will be scored from 0 (no consumption) to 3 (daily consumption) with a higher score indicating greater consumption of live bacteria. Consumption of vitamins and probiotics will be scored from 0 (no consumption) to 3 (daily consumption) with a higher score indicating greater consumption of vitamins and probiotics. Seven gastrointestinal symptoms will be scored from 0 (none) to extreme (4), with a maximum score of 28. A higher score indicates worse gastrointestinal symptoms.
Histopathology | intraoperative
  Synovial and tibial plateau samples will be collected intraoperatively and graded for synovitis. Intimal hyperplasia, sub-synovial infiltrate, fibrosis, fibrin deposition, perivascular edema, and vascularization will be graded on a scale of 0 (none) to 3 (severe). A higher score indicates greater synovial inflammation, with a total score range from 0 to 18.
Immunohistochemistry | intraoperative
  Synovial and tibial plateau samples will be collected intraoperatively, and the number of macrophages per mm² will be determined. A higher number indicates greater synovial inflammation.
Inflammatory Blood Marker: C-Reactive Protein | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of C-Reactive Protein (CRP) will be measured (mg/mL) and compared over time and between groups. Elevated CRP levels are an indicator of inflammation.
Inflammatory Blood Marker: Interleukin-1B | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of Interleukin-1B (IL-1β) will be measured (pg/mL) and compared over time and between groups. Elevated IL-1β levels are an indicator of inflammation.
Inflammatory Blood Marker: Interleukin-6 | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of Interleukin-6 (IL-6) will be measured (pg/mL) and compared over time and between groups. Elevated IL-6 levels are an indicator of inflammation.
Inflammatory Blood Marker: Interleukin-8 | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of Interleukin-8 (IL-8) will be measured (pg/mL) and compared over time and between groups. Elevated IL-8 levels are an indicator of inflammation.
Inflammatory Blood Marker: Tumor Necrosis Factor Alpha | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of Tumor Necrosis Factor Alpha (TNF-α) will be measured (pg/mL) and compared over time and between groups. Elevated TNF-α levels are an indicator of inflammation.
Inflammatory Blood Marker: Erythrocyte Sedimentation Rate | pre-operative, 6 weeks
  Participants will provide a blood sample. The Erythrocyte Sedimentation Rate (ESR) will be measured (mm/hr) and compared over time and between groups. Elevated ESR is an indicator of inflammation.
Inflammatory Blood Marker: Alkaline Phosphatase | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of Alkaline Phosphatase (ALP) will be measured (units/L) and compared over time and between groups. Elevated ALP levels can indicate inflammation, and may occur during periods of increased bone remodeling or tissue regeneration.
Inflammatory Blood Marker: Calcium | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of calcium will be measured (mmol/L) and compared over time and between groups. Lower calcium levels are an indicator of inflammation.
Inflammatory Blood Marker: Albumin | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of albumin will be measured (g/L) and compared over time and between groups. Decreased levels of albumin are often observed in conditions associated with inflammation.
Inflammatory Blood Marker: Urate | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of urate will be measured (μmol/L) and compared over time and between groups. Elevated urate levels are an indicator of inflammation.
Inflammatory Blood Marker: Total Protein | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of total protein will be measured (g/L) and compared over time and between groups. Elevated protein levels can indicate inflammation.
Inflammatory Blood Marker: Creatinine | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of creatinine will be measured (μmol/L) and compared over time and between groups. Elevated creatinine levels can indicate inflammation.
Inflammatory Blood Marker: Vitamin D | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of Vitamin D will be measured (nmol/L) and compared over time and between groups. Decreased Vitamin D levels are an indicator of inflammation.
Inflammatory Blood Marker: White Blood Cell Count | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of white blood cells (WBC) will be measured (cells/μL) and compared over time and between groups. Elevated WBC levels are an indicator of inflammation.
Inflammatory Blood Marker: Red Blood Cell Count | pre-operative, 6 weeks
  Participants will provide a blood sample. Levels of red blood cells (RBC) will be measured (cells/μL) and compared over time and between groups. Decreased RBC levels are an indicator of inflammation.
Inflammatory Blood Marker: Hemoglobin Concentration | pre-operative, 6 weeks
  Participants will provide a blood sample. Hemoglobin concentration (Hgb) will be measured (g/L) and compared over time and between groups. Decreased Hgb concentration is an indicator of inflammation.
Inflammatory Blood Marker: Hematocrit Percentage | pre-operative, 6 weeks
  Participants will provide a blood sample. Hematocrit (Hct) percentage will be measured (%) and compared over time and between groups. Decreased Hct percentage is an indicator of inflammation.
Inflammatory Blood Marker: Platelet Count | pre-operative, 6 weeks
  Participants will provide a blood sample. Platelet counts will be measured (cells/μL) and compared over time and between groups. Elevated platelet counts are an indicator of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanting, BESc, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No